CLINICAL TRIAL: NCT01066780
Title: Evaluation of the ClearVoice™ Strategy in Adults Using HiResolution® Fidelity 120® Sound Processing
Brief Title: ClearVoice Sound-processing Strategy for AB HiRes 120 Cochlear Implant Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Bionics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR0309
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2012-10

CONDITIONS: Implant
Keywords: cochlear implant; adults; HiResolution; Fidelity 120; listening benefits; noise; cochlear implant benefit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: ClearVoice Medium (Experimental): Chronic use of ClearVoice MEDIUM for two weeks followed by chronic use of ClearVoice HIGH for two weeks.
  Interventions: Device: ClearVoice
- Group B: ClearVoice High (Experimental): Chronic use of ClearVoice HIGH for two weeks followed by chronic use of ClearVoice MEDIUM for two weeks.
  Interventions: Device: ClearVoice

INTERVENTIONS:
Device: ClearVoice — ClearVoice is a sound processing strategy designed to improve listening ability in some challenging everyday listening environments for users of the Harmony® HiResolution® Bionic Ear System (Harmony®)

SUMMARY:
The purpose of this study is to collect information about how the new sound-processing affects the ability to hear in everyday listening situations.

ELIGIBILITY:
Inclusion Criteria:

* Post-lingually deafened,
* experienced (6 months device use),
* adult users of the Harmony HiResolution Bionic Ear System and HiRes Fidelity 120 sound processing.
* English language proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (9):
  - House Ear Clinic, Los Angeles, California
  - Carle Clinic Association, Urbana, Illinois
  - University of Kentucky, Lexington, Kentucky
  - The Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Midwest Ear Institute, Kansas City, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Nova Scotia Hearing and Speech Centres, Halifax, Nova Scotia
  - Sunnybrook Health Sciences Centre, Toronto

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were fit acutely at the Baseline Visit (Visit 1) with ClearVoice Low and underwent acute speech perception testing. Each subject was then randomized to Group A or Group B.
Groups:
- Group A: Received ClearVoice MEDIUM Followed by HIGH: Two weeks of chronic use of ClearVoice MEDIUM followed by two week of chronic use of ClearVoice HIGH.
- Group B: Received ClearVoice HIGH Followed by MEDIUM: Two week of chronic use of Clearvoice HIGH followed by two week of chronic use of ClearVoice MEDIUM.
Period: Overall Study
Arm/Group | Group A: Received ClearVoice MEDIUM Followed by HIGH | Group B: Received ClearVoice HIGH Followed by MEDIUM
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1
Not completed — Withdrawn prior to ClearVoice exposure. | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | ClearVoice
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (16.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Speech Perception of Standardized Sentences Presented From Recorded Format in Speech-spectrum Noise
Description: This was a within subjects design where scores on the AzBio sentence test in speech spectrum noise were compared against quiet scores at the 2-Week and 4-Week Follow-up Visit. The AzBio corpus of sentences consists of 33 lists of 20 sentences each (6 to 10 words per sentence) that have been equated for intelligibility. Two AzBio sentence lists were scored at each follow-up visit (2-Week and 4-Week) with either ClearVoice MEDIUM or ClearVoice HIGH enabled and averaged together. Two AzBio sentence lists were also administered in quiet at each visit. The ClearVoice score minus the quiet score provided the difference in score for the analysis.
Time Frame: 4 Weeks
Measure: Mean (Standard Deviation); unit: percentage of words scored correctly
Groups:
- Group 1: Primary efficacy analyses were based on data from the 46 subjects that completed the study.
Arm/Group | Group 1
Number analyzed (Participants) | 46
percentage of words scored correctly
  ClearVoice Setting Medium | 8.7 (10.10)
  ClearVoice Setting High | 10.6 (10.20)

2. Secondary Outcome: The AzBio Sentences Will be Administered in Recorded Format in Multi-talker Babble.
Time Frame: 2-4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days before submission for publication, presentation or use, Institution or Principal Investigator will submit to Sponsor for review and comment any proposed oral or written Publication. Sponsor will have the right to request any modification of any Publication if in Sponsor's reasonable opinion that Publication would jeopardize a patent application or patent.